CLINICAL TRIAL: NCT05257746
Title: Perioperative and Postoperative Evaluation of Rectal and Urogenital Function in Patients Undergoing Rectal Resection
Acronym: PERIFUNC
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: VTG-10
Record Dates: First submitted 2022-02-07; First posted 2022-02-25 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Rectal Surgery
MeSH Terms: interventions — Proctectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Rectal resection — Open or minimally invasive rectal resection with total mesorectal excision

SUMMARY:
The aim of this study is the systematic analysis of the development of perioperative rectal and urogenital function in patients undergoing rectal resection with total mesorectal excision and the identification of risk factors for urogenital and sphincter function loss after this procedure. Knowledge of the corresponding risk factors could enable the identification of patient cohorts that could benefit from an intensified or altered postoperative treatment path. The results of this study could thus significantly influence the clinical management of patients with rectal cancer and improve the functional outcome in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing rectal resection with total mesorectal excision

Exclusion Criteria:

* primary or secondary removal of rectal sphincter apparatus
* patients with enterostomy persisting 12 months after initial rectal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing rectal resection with total mesorectal excision
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of pelvic function before and after rectal resection | 5 years
  Rectal and urogenital function will be assessed preoperatively and 12-24 months and 5 years postoperatively using the PERIFUNC score questionnaire, resulting in a score between 0 and 120. Higher scores mean a worse outcome (worse pelvic function).
Rectal sphincter function before and after rectal resection | 5 years
  Sphincter function will be assessed by manometry preoperatively and 12 - 24 months and 5 years postoperatively
Assessment of stool continence before and after rectal resection | 5 years
  Stool continence will be assessed preoperatively and 12-24 months and 5 years postoperatively using the LARS score questionnaire, resulting in a score between 0 and 42. Higher scores mean a worse outcome (worse stool continence).

SECONDARY OUTCOMES:
Operating time [min] | during surgery
  Time from skin incision until placement of last skin staple/suture.
Intraoperative blood loss [mL] | during surgery
  Intraoperative blood loss presents the amount of blood lost from skin incision until skin closure. Spilling water and ascites will be subtracted. Swabs will be squeezed and their content will also be sucked and added to the fluid collected in the suction containers
Duration of postoperative hospital stay [days] | At day of discharge, assessed up to 90 days
  Postoperative day 1 until day of discharge
Duration of postoperative intermediate/intensive care unit stay [days] | At day of discharge, assessed up to 90 days
  Postoperative day 1 until day of discharge
Frequency of peri-operative morbidity after resection | 90 days after surgery
  Frequency of peri-operative complications after resection
Kind of peri-operative morbidity after resection | 90 days after surgery
  Kind of peri-operative complications after resection

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Fritzmann, Dr., Principal Investigator — Technical University Dresden
Locations (1):
- Department of Gastrointestinal-, Thoracic and Vascular Surgery University Hospital Carl Gustav Carus Technische Universität Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No
Following publication of study results, de-identified patient data will be made available upon reasonable request